CLINICAL TRIAL: NCT07083154
Title: Efficacy, Safety, and Tolerability of a GLP-1/GCG Dual Receptor Agonist in Type 2 Diabetes With Early Dementia: A Multicenter, Randomized, Parallel-group, Double-blind, Placebo-controlled Trial
Brief Title: GLP-1/GCG Dual Agonist in Type 2 Diabetes With Early Dementia (LIGHT-COG Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Nanjing First Hospital, Nanjing Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Xiangya Hospital of Central South University (Other); Huadong Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-0502-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Dementia, Mild; Mild Cognitive Impairment; Type 2 Diabetes
Keywords: Type 2 Diabetes; Mild Dementia; Mild Cognitive Impairment; GLP-1/GCG Dual Agonist; Cognitive Dysfunction; Early Dementia
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Cognitive Dysfunction; Diabetes Mellitus, Type 2 | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mazdutide group (Experimental): Participants will receive weekly subcutaneous injections of mazdutide (starting at 2.0 mg, with stepwise dose escalation to a target maintenance dose of 4.0 mg and optional adaptive increase to 6.0 mg if necessary and tolerated) , in addition to their existing glucose-lowering therapy.
  Interventions: Drug: Mazdutide
- Placebo group (Placebo Comparator): Participants will receive weekly subcutaneous injections of matched placebo, in addition to their existing glucose-lowering therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mazdutide — Mazdutide injection (pre-filled auto-injector pen) is administered subcutaneously at the same time each week. The starting dose is 2.0 mg administered once weekly (QW). Based on individual patient tolerance, the dose should be gradually increased to the target therapeutic dose of 4.0 mg QW over a period of 4 to 12 weeks. The protocol permits adaptive dose escalation up to 6.0 mg weekly when clinically indicated. For participants unable to tolerate dose increases, treatment continue at their maximum tolerated dose. The total intervention duration is 76 weeks.
  Other Names: IBI362
  Arms: Mazdutide group
Drug: Placebo — Placebo injection (pre-filled auto-injector pen) is administered subcutaneously at the same time each week. The starting dose is 2.0 mg administered once weekly (QW). Based on individual patient tolerance, the dose should be gradually increased to the target therapeutic dose of 4.0 mg QW over a period of 4 to 12 weeks. The protocol permits adaptive dose escalation up to 6.0 mg weekly when clinically indicated. For participants unable to tolerate dose increases, treatment continue at their maximum tolerated dose. The total intervention duration is 76 weeks.
  Arms: Placebo group

SUMMARY:
The LIGHT-COG study is a 76-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group clinical trial. A total of 420 type 2 diabetes patients with early dementia are randomized 1:1 to either the active treatment group (receiving subcutaneous injections of mazdutide weekly, with stepwise dose escalation to a maintenance dose per protocol) or the placebo group (receiving matched placebo injections). The primary objective is to evaluate the potential disease-modifying effects of mazdutide on cognitive dysfunction in type 2 diabetes.

DETAILED DESCRIPTION:
The LIGHT-COG study is a 76-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial investigating the potential disease-modifying effects of the GLP-1/GCG dual receptor agonist mazdutide on cognitive dysfunction in 420 patients with type 2 diabetes (T2D) and early dementia. Participants will be randomized 1:1 to receive either weekly subcutaneous injections of mazdutide (starting at 2.0 mg, with stepwise dose escalation to a target maintenance dose of 4.0 mg and optional adaptive increase to 6.0 mg if necessary and tolerated) or matched placebo, in addition to their existing glucose-lowering therapy. The primary objective is to assess cognitive improvement, with key secondary endpoints including brain structure and function alterations, metabolic improvement, neurodegenerative biomarkers, and safety outcomes.

Participants will undergo comprehensive cognitive and metabolic assessments at baseline, followed by safety visits at Week 4 and every 8 weeks thereafter for monitoring of adverse events, adherence, and metabolic parameters. Comprehensive evaluations at Weeks 28, 52, and 76 will include cognitive assessments, advanced neuroimaging, and metabolic profiling. During the study period, if a subject's study drug has been titrated to the maximum tolerated dose or the maximum protocol-specified dose (6 mg), and glycemic control remains suboptimal (fasting venous blood glucose or fingertip capillary blood glucose > 8.5 mmol/L on two consecutive measurements) during follow-up, individualized rescue therapy may be initiated upon the investigator's judgment. The choice of rescue regimen should be based on the investigator's comprehensive assessment of the subject's specific condition, including but not limited to glycemic levels, complications, hepatic and renal function, and risk of hypoglycemia. Optional rescue medications include insulin glargine, metformin, gliclazide modified-release, and acarbose. The investigator shall closely monitor the response to rescue therapy. The study should be terminated if any of the following occurs: inadequate glycemic control after rescue therapy, intolerance to rescue medications, or any other situation necessitating withdrawal as judged by the investigator. All decision-making basis, selection of rescue regimen, and efficacy evaluations must be thoroughly documented.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus (T2DM).
2. Aged 50-75 years (inclusive), male or female.
3. Early symptomatic dementia (Mild cognitive impairment or mild dementia), defined as:

   1. MMSE score >20 and <27,
   2. CDR global score 0.5-1.0 (inclusive), with a CDR memory subscore ≥0.5,
   3. Subjective memory complaints for ≥6 months.
4. Stable glycemic control regimen for ≥3 months prior to screening, meeting one of the following:

   1. Lifestyle/dietary intervention alone (no glucose-lowering drugs),
   2. Oral antidiabetic drugs (OADs), with or without once-daily basal insulin.
5. HbA1c 7.0-9.0% (inclusive) at screening.
6. BMI ≥20 kg/m², with stable weight (fluctuation <5%) for ≥3 months.
7. Stable treatment regimen for cognitive impairment for at least 3 months prior to screening and commit to its continuation throughout the study period, meeting one of the following criteria:

   1. No treatment: Not receiving any pharmacological or non-pharmacological interventions for cognitive impairment;
   2. Non-pharmacological therapy only: Engaged exclusively in non-drug interventions (e.g., cognitive training);
   3. Pharmacological therapy: Using approved symptomatic cognitive-enhancing medications (e.g., cholinesterase inhibitors, NMDA receptor antagonists), excluding disease-modifying therapies for Alzheimer's disease (AD).
8. Ability to comply with systematic cognitive and functional assessments.
9. Fully understands the trial protocol, voluntarily signs the informed consent form (ICF), and agrees to adhere to all study requirements and restrictions.

Exclusion Criteria:

1. Evidence of neurodegenerative disorders, including:

   1. Frontotemporal dementia (FTD) and its variants
   2. Parkinson's disease (PD), dementia with Lewy bodies (DLB)
   3. Progressive supranuclear palsy (PSP), corticobasal degeneration (CBD)
   4. Multiple system atrophy (MSA), multiple sclerosis (MS), Huntington's disease (HD)
2. With current or history of clinically significant psychiatric disorders within the past 2 years, including but not limited to: schizophrenia, bipolar disorder, major depressive disorder, generalized anxiety disorder, or personality disorders.
3. With a Patient Health Questionnaire-9 (PHQ-9) score ≥10 at screening, or a Generalized Anxiety Disorder Scale-7 (GAD-7) score ≥10 at screening.
4. History of stroke (ischemic/hemorrhagic), transient ischemic attack (TIA), or epileptic seizure within 3 months prior to screening; Current or prior diagnosis of central nervous system (CNS) disorders that may impair cognitive function, including but not limited to:

   CNS infections, Intracranial tumors, Metabolic encephalopathy, Neurological disorders due to malnutrition, or Severe traumatic brain injury.
5. Acute hyperglycemic/hypoglycemic events within 1 year, including: Diabetic ketoacidosis (DKA), hyperosmolar hyperglycemic state (HHS), and Hypoglycemic coma
6. Use of GLP-1R agonists, GLP-1R/GIPR dual agonists, or GLP-1R/GCGR dual agonists within 3 months prior to screening.
7. Regular use (>2 doses/week) of moderate-to-strong anticholinergic drugs within 4 weeks prior to screening; Use within 3 months prior to screening of: Anti-Parkinsonian drugs, Antiepileptic drugs, Antipsychotics, Morphine and opioid analgesics (Exemption: Short-term use [<5 days] for surgery/acute injury, if completed >4 weeks before screening); Use within 4 weeks prior to screening of: CNS stimulants; Medical/recreational cannabis, cannabinoids, or cannabidiol (CBD).a. Moderate/high anticholinergics, antiparkinsonian/antiepileptic drugs.
8. Alcohol abuse (defined as >21 units/week for men or >14 units/week for women; 1 unit = 360 mL beer, 150 mL wine, or 45 mL spirits).
9. Medical history of:

   1. Medullary thyroid carcinoma (MTC), pancreatitis
   2. Multiple endocrine neoplasia type 2 (MEN2)
   3. Gallbladder/biliary disease, severe gastrointestinal disorders, or bowel resection
   4. Active malignancy
10. Uncontrolled or potentially unstable diabetic retinopathy/maculopathy.
11. Severe organ dysfunction, including:

    1. ALT/AST >3× upper limit of normal (ULN)
    2. eGFR <45 mL/min/1.73m² (CKD-EPI equation)
    3. Unstable angina, myocardial infarction (MI), or NYHA Class II+ heart failure within 3 months
12. Known/suspected hypersensitivity to the investigational product or related compounds
13. Pregnancy, lactation, or women of childbearing potential not using highly effective contraception.
14. MRI contraindications (e.g., metal implants, claustrophobia).
15. Participation in other clinical trials within 3 months, involving an investigational medicinal product or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study.
16. Any other condition deemed by the investigator to compromise safety or interfere with study assessments.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-09-27 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Integrated Alzheimer's Disease Rating Scale (iADRS) Score Change | From Baseline to Week 28, 52 and 76
  The change in Integrated Alzheimer's Disease Rating Scale (iADRS) scores from baseline to Week 28, 52, and 76 will be compared between the treatment group and the placebo group to assess the drug's potential to improve or slow cognitive decline. iADRS is a composite endpoint that integrates cognitive and functional assessments (scores from Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) and Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living（ADCS-iADL）) to generate a total score (range: 0-144).
  The calculation formula is: iADRS score = (85 - ADAS-Cog13 score) + ADCS-iADL score
  A lower score indicates more severe cognitive and functional impairment.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) Score Change | From Baseline to Week 28, 52 and 76
  The change in Mini-Mental State Examination (MMSE) scores from baseline to Week 28, 52 and 76 will be compared between the treatment group and the placebo group to assess the drug's potential to improve or slow cognitive decline. It assesses multiple cognitive domains, including orientation, memory, attention and calculation, recall ability, language, and visuospatial skills. The total score ranges from 0 to 30, with higher scores indicating better cognitive function.
Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) Score Change | From Baseline to Week 28, 52 and 76
  The change in Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) scores from baseline to Week 28, 52 and 76 will be compared between the treatment group and the placebo group to assess the drug's potential to improve or slow cognitive decline. The score ranges from 0 to 18, with higher scores indicating greater severity of cognitive and functional impairment.
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) Score Change | From Baseline to Week 28, 52 and 76
  The change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) scores from baseline to Week 28, 52 and 76 will be compared between the treatment group and the placebo group to assess the drug's potential to improve or slow cognitive decline. The score ranges from 0 to 85, with higher scores indicating more significant cognitive impairment.
Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL) Score Change | From Baseline to Week 28, 52 and 76
  The change in Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL) scores from baseline to Week 28, 52 and 76 will be compared between the treatment group and the placebo group to assess the drug's potential to improve or slow functional decline. The total score ranges from 0 to 59, with lower scores indicating more severe functional impairment.
Change in Total Brain Volume | From Baseline to Week 76
  The change in total brain volume evaluated by structural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Total White Matter Volume | From Baseline to Week 76
  The change in total white matter volume evaluated by structural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Total Gray Matter Volume | From Baseline to Week 76
  The change in total gray matter volume evaluated by structural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Cerebrospinal Fluid Volume | From Baseline to Week 76
  The change in cerebrospinal fluid volume evaluated by structural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Total White Matter Lesion Volume | From Baseline to Week 76
  The change in total white matter lesion volume evaluated by sturctural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Cortical Gray Matter Lobar Volumes | From Baseline to Week 76
  The change in cortical gray matter lobar volumes evaluated by sturctural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Subcortical Nuclei Volumes | From Baseline to Week 76
  The change in subcortical nuclei volumes evaluated by stuctural MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Changes in MRI-derived Alzheimer's disease (AD) signature region volumes | From Baseline to Week 76
  The AD signature regions included hippocampus, parahippocampal, entorhinal, inferior parietal lobule, precuneus, and cuneus.
Changes in cortical thickness of AD-susceptible regions | From Baseline to Week 76
  The meta- regions of interest (ROI) mean cortical thickness measure was computed from 12 brain regions previously shown to differentiate between patients with AD and healthy controls:bilateral entorhinal cortex, inferior temporal, midtemporal, inferior parietal, fusiform, and precuneus regions.
Alterations in Resting-State Functional MRI-derived Brain Network Connectivity | From Baseline to Week 76
  The alterations in brain network functional connectivity (e.g. auditory network, visual network, default mode network, salience network, and sensorimotor network, etc.）evaluated by functional MRI from baseline to Week 76 will be compared between the treatment group and the placebo group.
Change in Blood-Based Neurodegeneration Biomarkers | From Baseline to Week 76
  The change in blood-based neurodegeneration biomarkers (includingAmyloid-β (Aβ42/40 ratio), Phosphorylated tau (p-tau217), Glial fibrillary acidic protein (GFAP), and Neurofilament light chain (NfL), etc.）evaluated by Simoa from baseline to Week 76 will be compared between the treatment group and the placebo group.
Rate of Progression from MCI to dementia | From Baseline to Week 76
  Difference in proportions of MCI patients progressing to dementia at Week 28, 52, and 76 (treatment vs. placebo).

OTHER OUTCOMES:
Incidence of Treatment-emergent Adverse Events | From Baseline to Week 76
  Difference in incidence of treatment-emergent adverse events during the trial period (treatment vs. placebo).
Incidence of Treatment-emergent Serious Adverse Events | From Baseline to Week 76
  Difference in incidence of serious adverse events during the trial period (treatment vs. placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, MD, PhD, Principal Investigator — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (7):
- China (7):
  - Department of Endocrinology, Xiangya Hospital of Central South University, Changsha, Hunan
  - Department of Endocrinology, Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Department of Endocrinology, Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Department of Endocrinology, Endocrine and Metabolic Disease Medical Center,Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu
  - Department of Endocrinology, Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Department of Endocrinology, Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Department of Endocrinology, Huadong Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Availability:
  De-identified participant data may be timely shared with qualified researchers upon request, subject to review and approval.
  Access Conditions:
  Data requests require a valid research proposal and signed data use agreement. Approval is contingent on compliance with applicable laws and ethical guidelines.
  Timing:
  Data will become available after study completion and primary publication for 3 years.
  Restrictions:
  Certain data types may be excluded due to privacy or regulatory requirements.
  Contact:
  Requests should be submitted to the study sponsor for consideration.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after study completion and primary publication for 3 years.
Access Criteria: Data requests require a valid research proposal and signed data use agreement. Approval is contingent on compliance with applicable laws and ethical guidelines.